CLINICAL TRIAL: NCT02991066
Title: Role of Microparticles in the Coagulopathy of Acute Promyelocytic Leukemia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 1309
Record Dates: First submitted 2016-03-02; First posted 2016-12-13 (Estimated); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Acute Promyelocytic Leukemia
Keywords: Acute promyelocytic leukemia; Coagulopathy; Microparticles; Mechanism
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute; Hemostatic Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood from patients with acute promyelocytic leukemia and from healthy volunteers is collected into 0.119M sodium citrate Vacuum tubes. platelet-free plasma is prepared within 4h using 2 serial centrifugations ( 15min at 1,500g, 2 min at 13,000g) and stored at -80℃ until use. A portion of PFP was filtered through a 0.1-um-pore size filter to collect microparticle-depleted plasma and stored at -80℃ until use. Experiments concerning procoagulant activity are detected immediately after blood collection.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients: patients with de novo acute promyelocytic leukemia with hemorrhage.
- Control: healthy volunteers.

SUMMARY:
Although the clinical application of differentiation therapy has made great success in the treatment of acute promyelocytic leukemia (APL), early fatal bleeding remains an unsolved problem which accounts for the main reason of induction failure in APL patients. The clinical manifestation of both serious bleeding and thrombosis illustrate the complexity of the pathogenesis of coagulopathy in APL. Despite extensive research, the pathogenesis of coagulopathy in APL is still unclear. Microparticles, 0.11μm in diameter, are small membrane vesicles released to circulation by blood cells and vascular endothelial cells during activation or apoptosis. Microparticles (MPs) derived from different cells types all exert procoagulant activity mediated by phosphatidylserine (PS) and carry some basic substances derived from their origin cells. Also, the biological activity of microparticles is often significantly higher than that of the cells they come from. According to these problems and background knowledge, our project aims to observe the roles of microparticles derived from APL cells and the procoagulant or profibrinolytic activating factors resided on these microparticles in the pathogenesis of coagulopathy in APL, and the effects of different induction therapies, chemotherapeutic drugs or differentiation agents on these microparticles and their procoagulant or profibrinolytic activating factors. To carry out this study, microparticles are obtained from patients who undergo different induction therapies at different time points or from primary bone marrow APL cells which are treated by different drugs in vitro at different time points, the expressions and activities of five procoagulant or profibrinolytic activating factors, which are highly expressed in APL cells, PS exposure and the functional state of these microparticles, will be dynamically monitored. Further study of the pathogenesis of coagulopathy in APL can provide clues and help for deep understanding of clinical manifestations, guiding clinical treatment as well as judging prognosis, and establishing theoretical basis for exploring new treatment.

DETAILED DESCRIPTION:
The investigators plan to measure routine laboratory parameters of coagulation and fibrinolysis, the procoagulant or profibrinolytic activity of microparticles (MPs), and explore the role of the procoagulant and profibrinolytic activating factor of MPs in the pathogenesis of coagulopathy in patients with APL.

i. Dynamic turbidimetry of plasma clot formation. The effects of MPs on the kinetics of fibrin formation and on the optical properties of clots are studied using dynamic turbidimetry of re-calcified plasma samples (platelet-free plasma and microparticle-depleted plasma) without adding any clotting activator. Clotting of plasma samples induced by Ca2+ is followed by monitoring the optical density at λ = 405 nm at 37 °C.

ii. Thrombin generation assay. The amount of thrombin formed in plasma upon re-calcification is measured directly using a modified thrombin generation test . Because fibrin interferes with colorimetric measurements, plasma samples are first defibrinated by adding reptilase followed by incubation at 37 °C. The clots are removed. Then a chromogenic substrate for thrombin is added to the plasma samples. Thrombin generation is started by adding CaCl2 with simultaneous recording of the absorbance at λ = 405 nm.

iii. Thrombin generating capacity of the MPs. MPs are reconstituted in defibrinated (reptilase treated), normal pooled microparticle-depleted plasma. Then a chromogenic substrate for thrombin is added to the samples. Thrombin generation is started by adding CaCl2 with simultaneous recording of the absorbance at λ = 405 nm.

iv. Thrombin generation inhibitory experiments. The following inhibitors are pre-incubated with the microparticles: Annexin V, anti-human tissue factor (TF) and irrelevant control immunoglobulin G (IgG). Then repeats the experiment iii.

v. Fibrinolytic activity. Incubate a fixed concentration of plasminogen with the plasma samples in the presence of a chromogenic substrate selective for plasmin. Plasmin formed from plasminogen bound at the surface of microparticles cleaves the chromogenic substrate and the released p-nitroaniline is detected by measuring A405nm as a function of time.

vi. Determination of fibrinolytic activity on microparticles. The capacity of microparticles to activate plasminogen is determined by incubating a fixed concentration of plasminogen (1mM) with the microparticles with or without t-PA and/or u-PA in the presence of a chromogenic substrate selective for plasmin. Plasmin formed from plasminogen bound at the surface of microparticles cleaves the chromogenic substrate and the released p-nitroaniline is detected by measuring A405nm.

vii. Fibrinolytic activity inhibitory experiments. The following inhibitors are pre-incubated with the microparticles: anti-human tissue type plasminogen activator (tPA) , anti-human urokinase type plasminogen activator (uPA), and respective irrelevant control IgGs; ε-aminocaproic acid and plasminogen activator inhibitor-1 (PAI-1).Then repeat the experiment vi.

ELIGIBILITY:
Inclusion Criteria:

* Patients with de novo APL accompanied by hemorrhage.
* The diagnosis was confirmed by the presence of t(15;17) and/or the PML (promyelocytic leukemia)/RARa(retinoic acid receptor alpha) fusion gene.
* Patients should receive single-agent arsenic trioxide (ATO) for induction therapy.

Exclusion Criteria:

* Patients with relapsed acute promyelocytic leukemia.
* Patients without evidence of bleeding.
* Patients younger than 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with acute promyelocytic leukemia
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2014-10; Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in the Levels and Cellular Origin of MPs at 5 Weeks | 5 weeks
  Demonstration that the some procoagulant or profibrinolytic activating factors expressed on MP in APL patients' plasma associate with the thrombin generating capacity and fibrinolytic activity of patients' plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Zhou, MD, PhD, Study Chair — First Affiliated Hospital of Harbin Medical University
Locations (1):
- the First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] de la Serna J, Montesinos P, Vellenga E, Rayon C, Parody R, Leon A, Esteve J, Bergua JM, Milone G, Deben G, Rivas C, Gonzalez M, Tormo M, Diaz-Mediavilla J, Gonzalez JD, Negri S, Amutio E, Brunet S, Lowenberg B, Sanz MA. Causes and prognostic factors of remission induction failure in patients with acute promyelocytic leukemia treated with all-trans retinoic acid and idarubicin. Blood. 2008 Apr 1;111(7):3395-402. doi: 10.1182/blood-2007-07-100669. Epub 2008 Jan 14. PMID 18195095
- [Background] Jacomo RH, Melo RA, Souto FR, de Mattos ER, de Oliveira CT, Fagundes EM, Bittencourt HN, Bittencourt RI, Bortolheiro TC, Paton EJ, Bendlin R, Ismael S, Chauffaille Mde L, Silva D, Pagnano KB, Ribeiro R, Rego EM. Clinical features and outcomes of 134 Brazilians with acute promyelocytic leukemia who received ATRA and anthracyclines. Haematologica. 2007 Oct;92(10):1431-2. doi: 10.3324/haematol.10874. PMID 18024380
- [Background] Dally N, Hoffman R, Haddad N, Sarig G, Rowe JM, Brenner B. Predictive factors of bleeding and thrombosis during induction therapy in acute promyelocytic leukemia-a single center experience in 34 patients. Thromb Res. 2005;116(2):109-14. doi: 10.1016/j.thromres.2004.11.001. Epub 2005 Jan 12. PMID 15907524
- [Background] Breccia M, Avvisati G, Latagliata R, Carmosino I, Guarini A, De Propris MS, Gentilini F, Petti MC, Cimino G, Mandelli F, Lo-Coco F. Occurrence of thrombotic events in acute promyelocytic leukemia correlates with consistent immunophenotypic and molecular features. Leukemia. 2007 Jan;21(1):79-83. doi: 10.1038/sj.leu.2404377. Epub 2006 Aug 24. PMID 16932337
- [Background] Tapiovaara H, Alitalo R, Stephens R, Myohanen H, Ruutu T, Vaheri A. Abundant urokinase activity on the surface of mononuclear cells from blood and bone marrow of acute leukemia patients. Blood. 1993 Aug 1;82(3):914-9. PMID 8338954
- [Background] Menell JS, Cesarman GM, Jacovina AT, McLaughlin MA, Lev EA, Hajjar KA. Annexin II and bleeding in acute promyelocytic leukemia. N Engl J Med. 1999 Apr 1;340(13):994-1004. doi: 10.1056/NEJM199904013401303. PMID 10099141
- [Background] Liu Y, Wang Z, Jiang M, Dai L, Zhang W, Wu D, Ruan C. The expression of annexin II and its role in the fibrinolytic activity in acute promyelocytic leukemia. Leuk Res. 2011 Jul;35(7):879-84. doi: 10.1016/j.leukres.2010.11.008. Epub 2010 Dec 10. PMID 21146216
- [Background] Sinauridze EI, Kireev DA, Popenko NY, Pichugin AV, Panteleev MA, Krymskaya OV, Ataullakhanov FI. Platelet microparticle membranes have 50- to 100-fold higher specific procoagulant activity than activated platelets. Thromb Haemost. 2007 Mar;97(3):425-34. PMID 17334510
- [Background] Bach RR. Tissue factor encryption. Arterioscler Thromb Vasc Biol. 2006 Mar;26(3):456-61. doi: 10.1161/01.ATV.0000202656.53964.04. Epub 2006 Jan 5. PMID 16397140
- [Background] Hron G, Kollars M, Weber H, Sagaster V, Quehenberger P, Eichinger S, Kyrle PA, Weltermann A. Tissue factor-positive microparticles: cellular origin and association with coagulation activation in patients with colorectal cancer. Thromb Haemost. 2007 Jan;97(1):119-23. PMID 17200778
- [Background] Tesselaar ME, Romijn FP, Van Der Linden IK, Prins FA, Bertina RM, Osanto S. Microparticle-associated tissue factor activity: a link between cancer and thrombosis? J Thromb Haemost. 2007 Mar;5(3):520-7. doi: 10.1111/j.1538-7836.2007.02369.x. Epub 2006 Dec 13. PMID 17166244
- [Background] Biro E, Sturk-Maquelin KN, Vogel GM, Meuleman DG, Smit MJ, Hack CE, Sturk A, Nieuwland R. Human cell-derived microparticles promote thrombus formation in vivo in a tissue factor-dependent manner. J Thromb Haemost. 2003 Dec;1(12):2561-8. doi: 10.1046/j.1538-7836.2003.00456.x. PMID 14738565
- [Background] Pereira J, Alfaro G, Goycoolea M, Quiroga T, Ocqueteau M, Massardo L, Perez C, Saez C, Panes O, Matus V, Mezzano D. Circulating platelet-derived microparticles in systemic lupus erythematosus. Association with increased thrombin generation and procoagulant state. Thromb Haemost. 2006 Jan;95(1):94-9. PMID 16543967
- [Background] Kwaan HC, Rego EM. Role of microparticles in the hemostatic dysfunction in acute promyelocytic leukemia. Semin Thromb Hemost. 2010 Nov;36(8):917-24. doi: 10.1055/s-0030-1267045. Epub 2010 Nov 3. PMID 21049391